CLINICAL TRIAL: NCT05076461
Title: Comparison of Ondansetron Versus Domperidone for Treating Vomiting in Acute Gastroenteritis in Children At a Resource Limited Setting
Brief Title: Ondansetron Versus Domperidone for Treating Vomiting in Acute Gastroenteritis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehsil Headquarter Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Tauseef Ahmad, Principal Investigator, Tehsil Headquarter Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TehsilHeadquarter
Record Dates: First submitted 2021-09-15; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Vomiting in Infants and/or Children; Acute Gastroenteritis
MeSH Terms: interventions — Ondansetron

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ondansetron group (Experimental): Children in ondansetron group received oral suspension of ondansetron as 0.15mg per body weight
  Interventions: Drug: Ondansetron
- Domperidone group (Experimental): Children in domperidone group, oral suspension of domperidone was given as 0.5 mg per kg body weight
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Ondansetron — Ondansetron group received oral suspension of ondansetron as 0.15mg per body weight

SUMMARY:
Most of the trials conducted comparing ondansetron and domperidone have been conducted among children aged below 5 or 6 years of age while no study from Pakistan has compared efficacy of these antiemetic agents among children up to 12 years of age. The findings of present study will give valuable evidence about the effectiveness of these antiemetic agents to prevent vomiting among children suffering with acute gastroenteritis at a resource limited setting of South Punjab, Pakistan.

DETAILED DESCRIPTION:
to compare the efficacy of ondansetron versus domperidone for treating vomiting in acute gastroenteritis in children at a resource limited emergency setting of South Punjab, Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Children of both genders aged below 12 years of age having 3 or more non-bilious, non-bloody vomiting episodes within 24 hours and with suggestive signs and symptoms of Acte Gastroenteritis.

Exclusion Criteria:

* Children who took any kinds of antiemetic in the last 6 hours of presentation of emergency department.
* Children having chronic liver disease, chronic kidney disease or congenital heart disease, neurological disorders, any kinds of malignancy, severe dehydration (requiring intravenous fluid replacement), severe acute malnutrition (weight-for-height below -3 standard deviation (SD) adopting WHO child growth protocols) or history known to allergy to antiemetics.

Ages: 1 Day to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Cessation of vomiting | 24 hours
  Children in ondansetron group received oral suspension of ondansetron as 0.15mg per body weight while in domperidone group, oral suspension of domperidone was given as 0.5 mg per kg body weight. Children in both study groups were administered designated drugs in the emergency department. Children were observed in the emergency department for 6-hours and discharged if they were vomiting free. All children were asked to follow up after 24 hours for the assessment of the effectiveness of the treatment for cessation of vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Tauseef Ahmad, MBBS, Principal Investigator — Tehsil Headquarter Hospital, Liaquatpur, Pakistan.
Locations (1):
- Tehsil Headquarter Hospital, Liaquatpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No